CLINICAL TRIAL: NCT03649516
Title: The Impact of Mobile APP Intervention ( iCKD APP) on Chronic Kidney Disease Care: A Multicenter, Randomized, Open, Controlled Trial
Brief Title: The Impact of Mobile APP Intervention ( iCKD APP) on Chronic Kidney Disease Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KMUHIRB-F(II)-20180055
Record Dates: First submitted 2018-08-07; First posted 2018-08-28 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2019-08

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: mHealth; Mobile application; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCKD APP Group (Experimental): Use iCKD APP
  Interventions: Device: iCKD APP
- Traditional Care Group (No Intervention): Accept traditional care

INTERVENTIONS:
Device: iCKD APP — Use iCKD APP to upload home bio-information data
  Arms: iCKD APP Group

SUMMARY:
* Apply Mobile APP Intervention ( iCKD APP) to current chronic kidney disease care program.
* Conduct a randomized clinical trial to evaluate the clinical effectiveness of this mobile device on health behavior improvement in chronic kidney disease patients.

DETAILED DESCRIPTION:
A mHealth app (iCKD APP) was designed to assist CKD patients to monitor their home bio-information data. Patients will be randomly assigned into the iCKD APP group(intervention) and traditional care group (control). Participants will be randomized into an 1:1 manner (intervention : control). Random assignment occurred after the consent and initial enrollment interview. Individuals randomized to the iCKD APP will provide with the equipment after randomization. Participants will follow for at least 6 months before the exit interview.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are 20 years old and above, Chinese speaking, and able and willing to provide informed consent.
* Subjects own mobile devices such as cell phones and tablets.
* Subjects were diagnosed with Chronic Kidney Diseases and were taking a single antihypertensive agent for more than three months or they are not receiving treatment but with systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg.

Exclusion Criteria:

* starting dialysis or having a kidney transplant (RRT)
* participating in other interventional study
* cognitively impaired
* unable to give consent
* life expectancy less than 1 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Compare clinics and home blood pressure | 3 months
  Systolic and diastolic blood pressure levels measured at both clinics and home will be compared between and within groups at various time points in study period.

SECONDARY OUTCOMES:
Achievement of Blood pressure control target | 3 months
  Achievement of Blood pressure control target will be compared between and within groups at various time points in study period.
The monitor rate of Home Blood pressure | 3 months
  The monitor rate of Blood pressure at home will be compared between and within groups at various time points in study period.

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Jyh Hwang, Study Chair — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No